CLINICAL TRIAL: NCT04779541
Title: National Survey Concerning Vaccination Against COVID-19 in Nursing Homes and Long-Term Care Units
Acronym: VACOVID-SENIOR
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-028; ar21-0004v0 (Other: research GDPR register)
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV-2; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — observation of the mechanisms of acceptance or rejection of the vaccine

SUMMARY:
The COVID-19 pandemic is a challenge for the French healthcare system, particularly among the elderly due to their particular vulnerability to the serious consequences of the disease, with an estimated mortality rate of around 30-35% among the frail elderly. The management of the health crisis could take a new turn in 2021 with the arrival in France of vaccines against the SARS-CoV-2 virus.

The objectives of this vaccination campaign are to reduce the morbi-mortality attributable to COVID-19 on the one hand, and to maintain essential activities related to the functioning of the country on the other hand and in particular the health system.

However, the distrust of vaccination, traditionally strong in France, could have a negative impact on this strategy. While the President of the Republic announced on November 24, 2020 that vaccination against SARS-CoV-2 would not be made compulsory, almost one French person in two declared in several surveys that they did not want to be vaccinated; the main criterion for acceptance of vaccination being advanced age (the older they are, the more French people declare accepting to be vaccinated).

In view of the gradual vaccine supply schedule for the year 2021, the French National Authority for Health established at the end of 2020 a prioritization by vaccine availability phases. The critical initial supply phase,which is currently taking place, is the one during which residents of retirement home and long-term care units are prioritized because of their particular vulnerability (age and co-morbidities) and their increased exposure to SARS-CoV-2.

For these reasons, and in order to carry out the current vaccination campaign in the most optimal way possible, this national survey is launching to evaluate the acceptance rate of the SARS-CoV-2 vaccine among people living in retirement homes and long-term care units, to understand the mechanisms of acceptance or rejection, and to draw up an initial large-scale inventory of the symptoms observed following vaccination.

ELIGIBILITY:
Inclusion Criteria:

* People aged 75 years and older in retirement homes or long-term care units who have accepted the SARS CoV-2 vaccine
* People aged 75 years and older in retirement homes or long-term care units who have refused the SARS CoV-2 vaccine
* National survey in france

Exclusion Criteria:

* Opposition of the elderly person and/or his or her relatives

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: all french seniors in retirement homes or long-term care units by SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Acceptance rate of the SARS-CoV-2 vaccine among people living in nursing homes and long-term care units | at baseline
  Number of acceptances of the vaccine with analysis of the reason for refusal.

SECONDARY OUTCOMES:
Symptoms related to vaccination against COVID-19 | at baseline
  description and identification of symptoms presented after vaccination of elderly patients

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France